CLINICAL TRIAL: NCT05250544
Title: The Effect of Stress Ball and Breathing Exercises on Fear and Pain in Adolescents Giving Polymerase Chain Reaction (rRT-PCR) Test
Brief Title: The Effect of Stress Ball and Breathing Exercises on Reducing Fear and Pain Associated with PCR Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayse Sonay Turkmen, Prof.Dr, Assoc.Prof., Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: stress ball-breathing exercise
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2022-11

CONDITIONS: Adolescent Behavior; Pain, Acute
Keywords: Adolescent; polymerase chain reaction; pain; afraid; stress ball; breathing exercise
MeSH Terms: conditions — Adolescent Behavior; Acute Pain; Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stress ball group (Experimental): For the adolescents in the stress ball group; Before the procedure, the adolescent's fear (with Childeren's Fear Scala (CFS)) will be evaluated and recorded by the adolescent, parent and observer. Then, the stress ball will be introduced to the adolescents and they will be asked to hold it in their desired hands. After explaining how to squeeze the stress ball, the PCR Test will start a few seconds after the adolescent starts to squeeze. As soon as the process starts, the stopwatch will be started, and when the process is finished, it will be stopped. When the PCR Test starts, the crying state of the adolescent will be observed and recorded. After the procedure, the adolescent's fear (Childiren's Fear Scala (CFS)) and pain (Wong Baker FACES) related to the procedure will be evaluated separately by the adolescent, parent and observer and recorded in the form.
  Interventions: Other: control group
- Breathin exercise group (Experimental): For the adolescents in the breathing exercise group; Before the procedure, the adolescent's fear (with Child's Fear Scala (CFS)) will be evaluated and recorded by the adolescent, parent and observer. Then, the breathing exercise will be introduced and applied to the adolescents. After explaining how to do the breathing exercise, the adolescent will be expected to complete the exercises. The PCR Test process will begin immediately after the exercise is complete. As soon as the process starts, the stopwatch will be started and will be stopped when the process is finished. After the procedure, the adolescent's fear (Childiren's Fear Scala (CFS)) and pain (Wong Baker FACES) related to the procedure will be evaluated separately by the adolescent, parent and observer and recorded in the form.
  Interventions: Other: control group

INTERVENTIONS:
Other: control group — For the adolescents in the control group; As soon as the process starts, the stopwatch will be started, and when the process is finished, it will be stopped. When the PCR Test starts, the crying state of the adolescent will be observed and recorded. After the procedure, the adolescent's fear (Childiren's Fear Scala (CFS)) and pain (Wong Baker FACES) related to the procedure will be evaluated separately by the adolescent, parent and observer and recorded in the form.

SUMMARY:
The COVID-19 pandemic continues to be one of the longest lasting pandemics experienced in recent times. Although the disease shows symptoms in different ways, the most effective diagnostic method known is the PCR test. This procedure is an unknown test method that many people have never had in their lifetime. Uncertainty in any subject causes stress and fear in the person. When the suspicion of a disease is added to this situation, the situation can reach even more serious dimensions. For this reason, it can be said that the PCR test can cause many problems, especially fear and pain. The most important health professional that the patient can reach before, during and after the test is the nurse. In order for the nurse to complete the test in a short time and with success, it may be necessary for the applicants to keep their fear levels under control and to support their fear management. In addition, the nurse plays an important role in the assessment and management of pain.

In the literature review, no study was found on reducing the fear and pain of the adolescents who gave the PCR Test. It is also thought that breathing exercises and stress ball can be an advantageous method in reducing pain and fear, considering their easy accessibility, affordable cost and long-term use. For this reason, this study was planned to determine the effect of stress ball and breathing exercises on the management of fear and pain that may occur due to PCR testing.

DETAILED DESCRIPTION:
Research type: Randomized controlled experimental study

Dependent variables: Adolescents' fear and pain levels from PCR testing Independent variables: Stress ball, breathing exercises, demographics

Hypotheses H0: Stress ball and breathing exercises have no effect on reducing fear and pain during the PCR test process.

H1: Stress ball has an effect on the level of fear that occurs during the PCR Test process.

H2: Breathing exercises have an effect on the level of fear that occurs during the PCR Test process.

H3: Stress ball has an effect on the level of pain that occurs during the PCR test process.

H4: Breathing exercises have an effect on the level of pain that occurs during the PCR test procedure.

The population of the study consists of adolescents aged 12-18 years who applied to Karaman Training and Research Hospital for PCR test. Power analysis was performed using the sample size G*Power (v3.1.9) program. The power of the study is expressed as 1-β (β = probability of type II error), and in general studies should have 80% power. Power analysis was performed to determine the adequacy of the sample size of the study; The power of the study was determined to be 0.95 with a significance level of 0.05, a confidence interval of 0.95, and an effect size of 0.97. Accordingly, there must be 29 people in each group. It was planned to carry out the research with a total of 96 children and their parents, 32 in each group, considering possible case losses during the research period.

Randomization The process of enrolling adolescents into groups will be randomly assigned. In the study, "stratification and block randomization methods" will be used in assigning participants to control and intervention groups. It has been reported in the literature that age, gender, and fear of interventional procedures are among the factors affecting the fear and stress experienced by children in interventional procedures. Accordingly, the children will be stratified as "girl and boy" for the gender variable, "afraid and not afraid" for the fear of the procedure, and randomization with blocks will be applied. The determined layers were created as codes obtained from the permutation-based computer program. At the beginning of the research, which letter would be the intervention or control group was determined by the closed opaque envelope method. Accordingly, the letter A will be used for the control group, B for the stress ball group, and C for the breathing exercise group. These block sets will be placed in envelopes of different colors and sizes by the researcher and kept in a black bag. It will be determined which stratum the children are in. It will be determined which group the determined child will be in according to the block set randomly drawn by the children from the black bag. If the next children are in the same layer, the block set will continue until the completion of the set. When it is determined that the incoming child is in a different layer, a new block set will be selected from the bag and the group will be determined.

Tabakalar Blok setler S1 Girl, Afraid CABC, BACC, BACB, ABAA, CACB, ACBB S2 Girl, Not afraid CACB, BCCC, ABBC, AACB, ABAC, ABAB S3 Man, Afraid ABBB, CBBC, CAAA, ABCC, ABCA, BCAC S4 Man, Not afraid CABC, BCAB, ACCB, ABAA, CACB, ACBB

Exclusion criteria from the study;

* Inability of the adolescents in the stress ball group to use the stress ball effectively throughout the procedure.
* Identification of extreme values that may affect the research data
* Child or parent's wish to leave the study

In data collection, Child and Parent Diagnosis Form, Children's Fear Scale (CFS), Wong Baker Faces Pain Scale (W-BFS), Stress ball and Breathing exercises applications will be used.

Child and Parent Identification Form It is a form prepared by the researcher by taking expert opinion and reviewing the literature to get information about the selected children and their parents for sampling. Form; It consists of questions that include the demographic characteristics of the child and his parents, whether the child has any disease, and the variables that may affect the child's pain and fear levels due to the procedure. Before starting the research, the interview and observation form will be applied to five children and their parents. Incomprehensible parts will be corrected and finalized. These children and their parents will be excluded from the research.

Children's Fear Scale (CFS) The CFS, which was first used in 2003, is a scale with proven validity and reliability developed to assess the child's fear level. Patients over the age of five can easily understand this method. There are five different facial expressions with no fear at one end of the scale and very intense fear at the other end, and are evaluated between 0-4 points. 0: no fear- 4: expresses extreme fear.

Wong Baker Faces Pain Comparison Scale (W-BFS) It is one of the most commonly used scales to measure the severity of pain in children. This scale was developed by Donna Lee Wong and Connie Morain Baker in 1981 and revised in 1983. The scale is used in the diagnosis of pain in children aged 3-18 years. It has been reported that the use of W-BPS is safe in children older than three years who can verbally express the degree of pain (Wong and Baker, 1988). There are face shapes and numbers on the scale. Pain is graded between "0" and "10" points. The level of pain felt is expressed with increasing degrees of facial expression . Ask the children "Which face shows your pain?", "How many points would you give your pain?" He will be asked to rate his pain by asking questions such as The parent will also be asked to evaluate the pain according to the child's reaction. Finally, the observer nurse will be asked to rate the pain she observes according to the child's reaction in another environment, without seeing the score given by the child and the parent. It has been stated that it is suitable for use in all cultures because it is a visual scale.

It has a plastic and soft structure that can be held comfortably. Each ball is about 7cm long and wide, it is a soft toy stuck in the hand, manipulated with fingers to relieve stress and muscle tension, exercise muscles. Contains no risk for children (not consisting of small parts that can be swallowed). The ball is in different colors such as orange, blue, green. Since all adolescents included in the study applied to the hospital with the suspicion of illness, in order to minimize the transmission of the disease by contact, separate balls will be given to all adolescents in the stress ball group and the balls will not be taken back.

Breathing Exercises Breathing exercises are applied for about 10 minutes and are mostly applied in the control of fear and stress. It has four different periods and each period lasts an average of four seconds. These periods are; breathing, waiting, breathing out and waiting periods. You can do this technique on proper breathing by following the steps below.

* Let's place our right hand on our chest and our left hand on our stomach.
* Let's breathe through our nose (counting to 4 inside us) wait for 4 seconds and breathe out slowly through our mouth (counting up to 4).
* If our rib cage (right hand) moves during breathing, it means we are breathing incorrectly.
* Let's just pay attention to the following while breathing: Our stomach will swell (left hand will move) when we breathe in, it will stay swollen as long as we hold our breath, and it will move inwards when exhaling.

In order for the adolescent to perform these applications correctly, instructions will be given by the researcher, and it will be ensured that they practice for about 10 minutes. In order to prevent the risk of contamination during breathing, the exercise will be done in a separate room, and the patient and the researcher will be masked. The room will be disinfected after each application.

Ethical and Legal Aspects of Research

In order to carry out the research, first of all, permissions were obtained from the authors, who made the Turkish validity and reliability of the scale to be used in the research, via e-mail. The aim of the study will be explained to the adolescents and their families who meet the research group selection criteria, their questions will be answered and their written consent will be obtained. It will be explained to the parents that the information they give will be kept confidential and will not be used anywhere else. In addition, those who do not want to participate in the study with verbal and written consent from the adolescents will not be included in the study. In the research, since the use of the human phenomenon requires the protection of individual rights, the relevant ethical principles "Informed Consent Principle", "Volunteering Principle" and "Principle of Protection of Confidentiality" will be fulfilled.

The data will be analyzed using descriptive statistics (percentage, mean, standard deviation, min-max value), difference analyzes (t-test in independent groups, paired t-test, mAnova, Mann Whitney U, Kruskal Walles), advanced analyzes when necessary (Tukey, Duncon etc.) and correlational analyzes (eg Pearson correlation analysis and Linear Regression analysis).

ELIGIBILITY:
Inclusion Criteria:

* The child is in the 12-18 age group,
* PCR Test was performed by the same nurse,
* The child has no pain (due to the disease, drug side effects, distension),
* The child does not have a hearing problem,
* PCR Test was performed in one go,
* The child has no history of epilepsy, migraine or vestibular disorders,
* Not taking analgesics in the last six hours,
* Absence of any medication that can affect the feeling of pain and fear that he uses constantly,
* The child and parent speak and understand Turkish comfortably,
* The child's mental development level to be able to answer the questions asked,
* Parents and children are willing to participate in the research,
* Obtaining written and verbal consent from parents.

Exclusion Criteria:

* Inability to perform PCR test in one go
* Presence of a chronic disease that may affect the sense of pain and fear of the adolescent.
* Having excessive fear and panic behavior before the procedure
* Negative effects on communication due to fear and panic behaviors
* Not being willing to participate in the study

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Fear score | 5 minutes
  Adolescents' fears will be evaluated (0-4 point)
Pain score | 5 minutes
  Adolescents' pain will be evaluated (0-4 point)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - KaramanogluMehmetbeyU, Karaman, Turkey
  - Karamanoglu Mehmetbey University, Karaman

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Apaydin Cirik V, Turkmen AS, Ayaz M. Effectiveness of stress ball and relaxation exercises on polymerase chain reaction (RRT-PCR) test-induced fear and pain in adolescents in Turkiye. J Pediatr Nurs. 2023 Jul-Aug;71:135-140. doi: 10.1016/j.pedn.2022.12.001. Epub 2022 Dec 14. PMID 36526480